CLINICAL TRIAL: NCT07371494
Title: SUPER-MINI PERCUTANEOUS NEPHROLITHOTOMY VERSUS FLEXIBLE URETEROSCOPY FOR RENAL STONES 20 MM OR LESS: A SINGLE-CENTER RANDOMIZED CONTROLLED TRIAL ASSESSING COST - ANALYSIS AND SAFETY IN NORTHERN VIETNAM
Brief Title: Super-Mini Percutaneous Nephrolithotomy Versus Flexible Ureteroscopy for Renal Stones ≤20 mm: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No. 876/GCN-HĐĐĐNCYSH-ĐHYHN
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Renal Calculi (Kidney Stones) ≤ 20 mm
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMP group (Experimental)
  Interventions: Procedure: Super-mini Percutaneous Nephrolithotomy
- fURS group (Experimental)
  Interventions: Procedure: Flexible Ureteroscopy

INTERVENTIONS:
Procedure: Super-mini Percutaneous Nephrolithotomy — Surgical removal of renal stones using super-mini PCNL technique
  Arms: SMP group
Procedure: Flexible Ureteroscopy — Endoscopic treatment of renal stones using flexible ureteroscope
  Arms: fURS group

SUMMARY:
Kidney stones measuring 20 mm or less are commonly managed using minimally invasive surgical techniques. Two widely used approaches are Super-mini Percutaneous Nephrolithotomy (SMP) and Flexible Ureteroscopy (fURS). Although both techniques are considered effective and safe, they differ in surgical approach, use of disposable equipment, postoperative recovery, and treatment cost. In resource-limited settings, economic considerations may play an important role in treatment selection.

This single-center randomized controlled trial was conducted at Bach Mai Hospital, Hanoi, Vietnam, to compare clinical outcomes, safety, and direct medical costs of SMP versus fURS in patients with renal stones ≤20 mm. Eligible patients were randomly assigned in a 1:1 ratio to undergo either SMP or fURS.

The primary outcome was the stone-free rate assessed by postoperative imaging. Secondary outcomes included operative time, postoperative complications, length of hospital stay, hemoglobin drop, and total direct treatment cost per case. The results of this study aim to provide evidence to support clinical decision-making for the management of renal stones, particularly in healthcare settings with limited resources.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years of age).
* Patients with renal stones measuring ≤20 mm in maximal diameter on preoperative imaging.
* No prior surgical or interventional procedure during the same hospital admission.
* Ability and willingness to provide written informed consent.

Exclusion Criteria:

* Pregnancy.
* Coagulation disorders or bleeding diathesis contraindicating surgery.
* Contraindications to either Super-mini Percutaneous Nephrolithotomy (SMP) or Flexible Ureteroscopy (fURS).
* Patients undergoing SMP or fURS for ureteral stones that migrated back into the kidney.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Stone-free rate (SFR) | 1 month after surgery
  Stone-free rate was defined as the absence of residual stone fragments >4 mm in maximal diameter on postoperative imaging. Stone-free status was assessed using plain abdominal radiography (KUB) on postoperative day 1 and non-contrast computed tomography (CT) at 1 month after surgery. The stone-free rate was determined based on the 1-month CT findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Bach Mai Hospital, Department of Urology, Hanoi, Vietnam